CLINICAL TRIAL: NCT02442154
Title: EARLY TRACHEOSTOMY VERSUS STANDARD OF CARE, A RANDOMIZED CONTROLLED CLINICAL TRIAL IN PATIENTS WITH SEVERE HEAD INJURY IN MULAGO HOSPITAL
Brief Title: Early Tracheostomy Versus Standard of Care in Patients With Severe Head Injury
Acronym: E-Trac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/HD07/2134U
Record Dates: First submitted 2015-04-29; First posted 2015-05-13 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2015-08

CONDITIONS: Severe Head Injury
Keywords: early tracheostomy; severe head injury; endotracheal intubation
MeSH Terms: conditions — Craniocerebral Trauma | interventions — Tracheostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early tracheostomy (Experimental): To do an early tracheostomy within 24hours of admission of the severely head injured patients
  Interventions: Procedure: Tracheostomy
- standard of care (No Intervention): To use the standard of care of mulago hospital for the management of the severely head injured patients

INTERVENTIONS:
Procedure: Tracheostomy — It is a surgical procedure which involves making an incision on the anterior aspect of the neck and opening a direct airway through an incision in the trachea with stitching the trachea to the skin and placement of a tube
  Arms: Early tracheostomy

SUMMARY:
Severe head injury is associated with airway compromise and poor respiratory effort. In Mulago Hospital intubation is the mainstay intervention and then patients are subjected to the wait and see strategy of delayed or no tracheostomy, very few undergo early tracheostomy, and some patients are left without an artificial airway.Using endotracheal tubes is associated with complications which have been shown to increase intensive care unit (ICU) and hospital stay, morbidity and mortality.

Tracheostomy has been reported to have advantages over translaryngeal intubation but the optimal timing of tracheostomy in patients with severe head injury is controversial. Studies done elsewhere have showed that patients with severe head injury who undergo early tracheostomy have better survival outcomes but no studies have been done in our setting

DETAILED DESCRIPTION:
Introduction; Most patients with severe head injury cannot protect their airway, have excessive secretions and inadequate spontaneous breathing which contributes to cerebral hypoxia. Thus, in their initial management the airway is secured with either an endotracheal tube (ETT) or a tracheostomy. In Mulago Hospital some of these patients are intubated and then subjected to the wait and see strategy of delayed or no tracheostomy, very few undergo early tracheostomy, and some patients are left without an artificial airway. Tracheostomy has been reported to have advantages over translaryngeal intubation but the optimal timing of tracheostomy in patients with severe head injury is controversial. Studies done elsewhere have showed that patients with severe head injury who undergo early tracheostomy have better outcomes.

Problem statement; Mulago hospital receives the largest number of patients with severe head injured with a mortality rate of 69%. Securing these patients airway using ETT is associated with complications which have been shown to increase ICU and hospital stay, morbidity and mortality. Furthermore, most intubated patients often require ICU admission for care of ETT and mechanical ventilation and yet these patients require little or no assistance from mechanical ventilation if the airway has been secured with a tracheostomy. With limited number of ventilators and beds in ICU and increased demand for ICU admission in Mulago hospital, this poses a challenge.

Objective; To compare 30 day mortality of severe head injured patients undergoing early tracheostomy versus standard of care in Mulago Hospital and the associated factors

Methodology; Randomized controlled clinical trial, open label, to be carried out in Mulago Hospital Trauma Centre, casualty, ICU, and neuro-surgical ward high dependence unit (3AHDU).

All patients above 10years with severe traumatic brain injury who meet the study criteria will be recruited and randomly assigned to either arm.

The patients on the early tracheostomy arm will undergo tracheostomy, done by an Otolaryngologist (ENT surgeon) or resident within 24 hours of admission, then admitted either in trauma center, ICU if there is space available, or Neurosurgery ward HDU. Patients will then receive routine care for the severe head injured patients as per Mulago hospital standards.

On the other arm the patients will receive the standard of care as per the attending clinician, and these are also admitted either in trauma Centre, ICU or Neurosurgery ward HDU where they also receive routine care for severe head injured patients as per Mulago hospital standards.

Follow up the primary outcome is 30day mortality The patients on both arms will be followed up for a maximum of 30 days To assess for; Acute complications of the tracheostomy (bleeding, subcutaneous emphysema, pneumothorax) Number of days on the mechanical ventilator and development of ventilator associated pneumonia (VAP) for the mechanically ventilated patients using; increase in respiratory rate, FiO2, temperature and White blood cell count from the baseline, consistency of the tracheal aspirate and culture of the tracheal aspirate.

Number of days patient requires sedation for the sedated patients. Length of ICU and hospital stay and glasgow coma scale (GCS) at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 10years
* GCS ≤ 8

Exclusion Criteria:

* Patients who undergo tracheostomies within 24hours of admission before randomization

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
30day mortality | within 30 days of follow up
  the number of deaths recorded within 30days of admission

SECONDARY OUTCOMES:
length of ICU and hospital stay | 30 days
  number of days spent in the ICU and hospital
incidence of ventilator associated pneumonia | 30days
  Number of days on the mechanical ventilator and development of VAP for the mechanically ventilated patients using; increase in respiratory rate, Fraction of inspired oxygen (FiO2), temperature and White blood cell count from the baseline, consistency of the tracheal aspirate and culture of the tracheal aspirate
duration of sedation | 30days
  number of days the patient receives sedatives
Glasgow coma scale on discharge | 30days
  level of consciousness on discharge

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Kwizera, Mmed, Study Director — Makerere Univervisity college of health science; Juliet Nalwoga, MBChB, Principal Investigator — Makerere University college of health science
Locations (1):
- Mulago Hospital Complex, Kampala, Kampala, Uganda